CLINICAL TRIAL: NCT03120312
Title: Short Term and Long Term Outcome for Elderly Patients Treated With Total Hip Replacements During Past 5 Years :A Retrospective Analysis
Brief Title: Short Term and Long Term Outcome for Elderly Patients Treated With Total Hip Replacement
Acronym: THR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, Professor, Second Hospital of Shanxi Medical University
Other Study IDs: ZGuo
Record Dates: First submitted 2017-04-15; First posted 2017-04-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Total Hip Replacement
Keywords: outcome
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: total hip replacement — primary hip replacement patients during past 5 years．

SUMMARY:
The is a retrospective analysis to study the characteristics of elderly patients treated with total hip replacements during past 5 years．

DETAILED DESCRIPTION:
Patients underwent total hip replacement due to removal of the hip caused by retrogressive lesions, is conducive to the improvement of hip function .But at the same time,the complications from patients accepted total hip replacement surgery will directly or indirectly affect the prognosis of the patients, resulting in patients with delayed recovery and increase the hospitalization time and cost. Serious complications can lead to patients deaths during perioperative period. This study was designed to provide a retrospective analysis of postoperative recovery, quality of life, and complications in patients undergoing hip replacement over the past five years, providing data for clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅱ-Ⅲ,elective operation patients，
2. NO other severe complication history

Exclusion Criteria:

1. Having severe comorbidity
2. not for the first time of joint replacement
3. Suffered from neurologic disorder or impaired mental state

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From January 2012 to July 30，2017，approximately 1500 cases of primary hip replacement in this study，including male ，female and bilateral replacements．
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life during 5 years after surgery | 5 years
  evaluate the quality of life after surgery by WHO QOL-BREF scale with interview ，WHO QOL-BREF scale includes five aspects: physical, psychological, social, environmental, integrated, divided into five levels

SECONDARY OUTCOMES:
The incidence of postoperative complications | from 7 days to 1 year
  Participants will be followed for the incidence of postoperative complications
Mortality during 5 years after surgery | during 5 years
  Participants will be followed for Survival rate during 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Guo, Study Chair — Second Hospital of Shanxi Medical University
Locations (1):
- Zheng Guo, Taiyuan, Shanxi, China

REFERENCES:
- [Background] Penrod JD, Litke A, Hawkes WG, Magaziner J, Doucette JT, Koval KJ, Silberzweig SB, Egol KA, Siu AL. The association of race, gender, and comorbidity with mortality and function after hip fracture. J Gerontol A Biol Sci Med Sci. 2008 Aug;63(8):867-72. doi: 10.1093/gerona/63.8.867. PMID 18772476
- [Background] Foss NB, Palm H, Krasheninnikoff M, Kehlet H, Gebuhr P. Impact of surgical complications on length of stay after hip fracture surgery. Injury. 2007 Jul;38(7):780-4. doi: 10.1016/j.injury.2006.08.028. Epub 2006 Oct 19. PMID 17054955
- [Background] Singh JA, Jensen MR, Harmsen WS, Gabriel SE, Lewallen DG. Cardiac and thromboembolic complications and mortality in patients undergoing total hip and total knee arthroplasty. Ann Rheum Dis. 2011 Dec;70(12):2082-8. doi: 10.1136/ard.2010.148726. Epub 2011 Oct 21. PMID 22021865
- [Background] Krecisz B, Kiec-Swierczynska M, Chomiczewska-Skora D. Allergy to orthopedic metal implants - a prospective study. Int J Occup Med Environ Health. 2012 Sep;25(4):463-9. doi: 10.2478/S13382-012-0029-3. Epub 2012 Dec 3. PMID 23212287
- [Background] Deutman R, Mulder TJ, Brian R, Nater JP. Metal sensitivity before and after total hip arthroplasty. J Bone Joint Surg Am. 1977 Oct;59(7):862-5. PMID 908716